CLINICAL TRIAL: NCT01319383
Title: A Phase I/II Investigation of the Effect of Vorinostat (VOR) on HIV RNA Expression in the Resting CD4+ T Cells of HIV-Infected Patients Receiving Stable Antiretroviral Therapy
Brief Title: The Effect of Vorinostat on HIV RNA Expression in the Resting CD4+ T Cells of HIV+ Pts on Stable ART
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Merck Sharp & Dohme LLC (Industry); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CID 0807; 1U01AI095052-01 (NIH)
Record Dates: First submitted 2011-03-17; First posted 2011-03-21 (Estimated); Results first posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-04

CONDITIONS: HIV-1 Infection
Keywords: HIV-1 Infection; HIV RNA <50 copies/mL; Stable ART; Resting CD4+ T cells; Leukapheresis; Vorinostat; HIV RNA expression; PK visits
MeSH Terms: interventions — Vorinostat

STUDY DESIGN:
Intervention Model Description: All participants eligible for study received the same open label drug
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open Label, Translational Research (Experimental): Vorinostat will be administered to all eligible participants in each step of each phase (period) of the study
  Interventions: Drug: Vorinostat

INTERVENTIONS:
Drug: Vorinostat — Vorinostat (VOR) 400mg will be given as single doses by mouth. Participants eligible to advance in study will have opportunity to receive more than one dose of VOR. Each participant will only take one dose of VOR in a 24 hour period. Repeat doses will be administered at least 24 hours apart, with option for dosing at intervals up to 96 hour
  Other Names: Zolinza; SAHA, or MK-0683; VOR

SUMMARY:
The purpose of this study is to compare HIV RNA expression and infection within resting (CD4)+ cells in HIV-infected patients on stable ART before and after a single exposure to Vorinostat (VOR), after exposure to short intervals of VOR, and after repeated short interval exposure to VOR dosed over several weeks.

Hypotheses:

1. The frequency of resting CD4+ T cell- associated HIV RNA (RCVL) will be increased following single and repeated exposure to VOR when given at appropriate intervals, and
2. That repeated exposure to VOR will reduce the frequency of HIV infection within resting CD4+ T cells (RCI)

DETAILED DESCRIPTION:
This is a Phase I-II single-center study in participants (ppts) with HIV-1 infection receiving stable ART, with plasma HIV RNA < 50 copies/mL. Baseline ART will be maintained throughout the study. Participants will be screened for study entry, and then undergo an initial leukapheresis evaluation at study entry to obtain resting CD4+ T cells for quantitation of resting CD4+ T cell infection (RCI) and resting CD4+ T cell- associated HIV RNA (RCVL) at a baseline evaluation. All 1st time leukapheresis participants, and others as requested based on prior latent pool determinations, will have HIV-1 DNA PCR done. All participants who enter the study will receive VOR at assigned study visits, and undergo repeat leukapheresis to measure the effects of VOR exposure.

Period One - Single and Multiple Dose Vorinostat (protocol versions (v) 3.0 and 5.0)

After signing the informed consent, completing screening and meeting all eligibility requirements, participants are enrolled and undergo a baseline leukapheresis (Visit 2). Participants exhibiting or not exhibiting a response [quantitation of resting CD4+ T cell infection (RCI) and resting CD4+ T cell- associated HIV RNA (RCVL)] to an ex vivo exposure to VOR will be evaluated for an in vivo response to a single dose of VOR 400 mg. Additionally participants complete a modified 24 hour pharmacokinetics (PK) analysis. All are monitored for adverse events (AEs) especially those that are dose-limiting. Safety monitoring included clinical labs, physical exams and assessment of medications and the onset of new signs and symptoms at all study visits.

Participants demonstrating in vivo a significant increase in the resting CD4+ T cell- associated HIV RNA (RCVL) after the single dose of VOR (protocol v3.0 and v5.0) are eligible to advance into Step 2. In Step 2 (protocol v5.0), participants are administered multiple doses of VOR. Each participant receives 22 total doses of VOR via 2 cycles of 11 doses each. Each cycle is 4 weeks in length. VOR 400 mg is administered on Monday, Tuesday and Wednesday followed by 4 days of no drug during the 1st 3 weeks. The 4th week of the cycle will have VOR administered on Monday and Tuesday, followed by a leukapheresis approximately 4 hours after the 11th dose (estimated peak drug level). Participants will be monitored throughout the 4 weeks for safety which includes the documentation of AEs, especially dose-limiting AEs, and other AEs associated with study procedures and events. After a rest period (approximately 5 - 8 weeks), participants repeat the 4 week cycle. Each cycle is analyzed for significant increase in resting CD4+ T cell- associated HIV RNA (RCVL) as compared to baseline (ex-vivo) and step 1 (single dose in-vivo) responses.

Period Two - Single, Paired Interval and Multiple Interval Doses of VOR (protocol v6.0)

Step 1: Enrollment into this study period was similar to the procedures in Period 1. Participants were consented to protocol v6.0, completed screening and after meeting eligibility, enrolled on the study at Visit 2. The leukapheresis, scheduled for Visit 2, was optional based on prior ascertainment of baseline parameters. Omission of this leukapheresis was determined by study PI, after analysis of lab data from previous leukapheresis procedures. Regardless of the completion of the leukapheresis procedure at Visit 2, study enrollment and collection of required research assays was completed at Visit 2. Participant were screened and enrolled into Step 1 until 12 evaluable participants successfully completed the multiple doses of VOR (Step 4), or until the study-stopping rules are met. It is estimated that up to 30 eligible participants may be screened and enrolled to provide a total of 12 evaluable participants who complete Step 3.

Step 2 included several visits: administration of VOR (visit 3), modified/abbreviated 8 hour PK analysis, leukapheresis procedure and safety follow up (Visit 4). After assessment and ascertainment of safe to proceed clinical status, each participant receive a single dose of VOR 400 mg. Participant remained in the clinic for observation and the collection of samples for the abbreviated PK. Four hours after the dose, the leukapheresis procedure was initiated. It was anticipated that the completion of Step 1 and 2 would occur over a minimum of 8 weeks. All participants must complete Step 2 prior to moving to Step 3. All participants are assessed after the Visit 3 leukapheresis for an in vivo response to the 400 mg of VOR.

Progression from Step 2 (single dose) to Step 3 (paired doses) was based on each participant's increase in RCVL following their first dose of 400 mg VOR (Visit 3), compared to that measured at baseline (Visit 2). Progression from Step 3 (paired doses) to Step 4 (multiple doses) will be based on each participant's increase in RCVL following the 2nd in a paired dose VOR 400 mg (total doses = 3, Visit 6), compared to that measured at baseline (Visit 2).

The goal of protocol v6.0 is to determine the optimal interval between two doses of VOR (Step 2), and the response of RCI (and secondarily RCLV) to repeated doses at this interval (Step 3).

Step 3 will be initiated at least 4 weeks after the completion of the Step 2 safety follow up visit (Visit 4). If greater than 60 days elapse between Visit 4 and Visit 5, participants will repeat screening Visit labs to qualify for continued study participation. In Step 3, two paired doses of VOR 400 mg will be administered. The interval between the 2 paired doses can be as short as 48 hours (2 days), and as much as 96 hours (4 days) apart from each other. Participants were assessed for in vivo response via a 3rd leukapheresis after the second of the paired doses of 400 mg VOR. The first three (3) participants will first be assessed for an in-vivo response after the 2nd dose of the paired doses given 48 hours (2 days) apart. Subsequent participants will be assessed for responses to paired doses separated by 48 hours, or the interval may be lengthened to as much 96 hours (4 days), as dictated by the accumulated responses observed in subsequent participants.

If at least 2 of the 3 participants with 48-hour intervals respond (defined as a significant within-subject increase in cell-associated HIV RNA), then 3 subsequent participants will receive 48-hour intervals. If 2 of these 3 respond (4 of 6 total), then 3 additional participants will receive 48-hour intervals. If among the first 6 evaluable participants receiving 48-hour intervals there are 3 non-responders, then subsequent participants will receive 72-hour intervals. Participants receiving 72-hour intervals will then be assessed in the same way as those receiving 48-hour intervals, to either continue additional participants at 72-hour intervals or to increase to 96-hour intervals. Step 3 will enroll until a total of 12 evaluable subjects with a measureable increase in cell-associated HIV RNA are obtained, and these participants have advanced to Step 4.

Our preliminary results from protocol version 5.0 (period 1) are consistent with the hypothesis that the complex cellular effects of HDAC inhibitor exposure require more than 24 hours to resolve. We observed what appears to be an antagonistic effect where a VOR dose blunts the effect of the next dose when two doses are given within 24 hours of each other. The purpose of Step 3 is to establish the optimal dosing interval in which a response to Vorinostat is sustained. Step 3 will study dosing intervals; starting with a 48-hour interval and moving to longer intervals between doses depending on the effect observed with the ultimate goal to determine the shortest interval that yields an optimal effect of VOR.

If a participant fails to respond in their initial Step 3 dosing interval, they can be eligible to repeat Step 3. They can re-enter or repeat Step 3 one time only. They will only re-enter Step 3 to test a longer dosing interval. Again, if > 60 days elapses between the final safety visit of step 3 (Visit 7) and their re-entry to Step 3, they will re-screen (visit 1 only) to qualify to continue in the study.

Step 4: After a period of at least 6 weeks, to allow data analysis, participants who demonstrate an in vivo response to the 2nd of the paired dose of VOR will proceed to Step 4 and receive 10 doses of VOR 400 mg administered at the same interval at which cell-associated HIV-RNA induction was observed in Step 3. If greater than 60 days elapse between Visit 7 and Visit 8, participants will repeat the screening visit labs to qualify for continued participation in the study. At the completion of 10 doses, participants will then be assessed via a 4th and final leukapheresis for in vivo response to the serial dosing of VOR.

It is anticipated that Step 4 will occur over a minimum of 4 weeks; however this may vary among participants based on their Step 3 dosing interval stage. Accumulated blood volumes and the timing between leukapheresis procedures will determine the length of time between each step. Participants completing this protocol (version 6.0), who respond initially in Step 3 will receive a total of 5200 mg of Vorinostat. Participant completing the study, who repeat Step 3, will receive a total of 6000 mg of Vorinostat. For reference, participants who completed the previous version (5.0) received a total of 10,000 mg of Vorinostat without clear evidence of any durable drug-associated toxicity thus far.

The change in the frequency of HIV-1 infection per million resting CD4 + cells will be measured after repeated short interval dosing with VOR in Step 4. The 4th leukapheresis (Visit 12) will be compared to the baseline leukapheresis done at Visit 2. If the VOR 400 mg dosing in Step 4 is interrupted due to toxicity or intolerance, then the leukapheresis will be performed as soon as possible after the VOR interruption. This is justified as if a depletion of resting cell infection can occur; new resting cell infection is unlikely to occur in the presence of ART. Test dosing in this Step will continue until the study's stopping (lack of response in five) or toxicity rules are met.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infection
2. Men, women age ≥18 years.
3. Ability, willingness to give written informed consent.
4. Able, willing to provide adequate locator information.
5. Karnofsky performance status >70.
6. Able, willing to adhere to therapy and adherent to ART.
7. Able,willing to comply with time requirements for study visits and evaluations.
8. On potent ART, defined as at least 2 nucleoside/nucleotide reverse transcriptase inhibitors plus a non-nucleoside reverse transcriptase inhibitor, integrase inhibitor, or a protease inhibitor without interruption (defined as missing doses for more than two consecutive days or more than four cumulative days) in the 24 weeks immediately prior to entry. Other potent fully suppressive antiretroviral combinations will be considered on a case-by-case basis. Prior changes in or elimination of medications for easier dosing schedule, intolerance, or other reasons are permitted if an alternative suppression regimen was maintained.
9. Adequate vascular access for leukapheresis.
10. Able to swallow pills without difficulty.
11. On combination ART for ≥ 18 months prior to study entry, no consecutive HIV-1 RNA values >50 copies/mL in that time period
12. CD4 cell count ≥ 300 cells/µl at screening.
13. All male study volunteers must agree not to participate in a conception process.
14. Must be seronegative for Hep C RNA, Hep B sAg within 90 days of entry
15. Must have adequate organ function as indicated by the following lab values:

Hematological: Absolute Neutrophil Count (ANC) ≥ 1,500/mcL Platelets ≥ 125,000/mcL Hgb ≥ 12 g/dL

Coagulation: Prothrombin Time or International Normalized Ratio (INR) ≤ 1.5x upper limit of normal (ULN)

Chemistry: K+ levels Within normal limits Mg++ levels > Lower limits of normal (LLN) but <1.5 x ULN Glucose Screening serum glucose(fasting/non-fasting) below 120 mg/dl.

Renal: Serum creatinine/calculated creatinine clearance* ≤ 1.3 X ULN OR ≥ 60 mL/min for participants with creatinine levels > 1.3 X ULN

Hepatic: Serum total bilirubin Total bilirubin < 1.5 times ULN. If total bilirubin is elevated, direct bilirubin will be measured and the participant will be eligible if the direct bilirubin is < 2 X ULN.

Aspartate amino transferase (AST) (SGOT) and Alanine amino transferase (ALT) (SGPT)≤ 2.0 X ULN Lipase <1.6 X ULN Alkaline Phosphatase ≤ 2.5 X ULN

*Creatinine clearance should be calculated per institutional standard.

Exclusion Criteria:

1. Received blood transfusions or hematopoetic growth factors within 90 days.
2. All women unless there is written documentation of menopause (absence of a period for ≥ one year), hysterectomy, oophorectomy, or tubal ligation.
3. The study PI is unable to construct a fully active alternative regimen based on previous resistance testing and/or treatment history
4. Use of atazanavir and raltegravir in background antiretroviral regimens.
5. Any antiretroviral medications that cannot be co-administered with Vorinostat within the 4 weeks of the first Vorinostat dose and anytime thereafter while on study.
6. Use of any of the following within 90 days prior to entry: systemic cytotoxic chemotherapy; investigational agents; immunomodulators (colony-stimulating factors, growth factors, systemic corticosteroids, HIV vaccines, immune globulin, interleukins, interferons); coumadin, warfarin, or other Coumadin derivative anticoagulants.
7. Any serious illness requiring systemic treatment or hospitalization, the subject must either complete therapy or be clinically stable on therapy, in the opinion of the site investigator, for at least 90 days prior to entry.
8. Compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric illness or a physical illness, e.g., infectious disease. Prisoner recruitment and participation is not permitted.
9. Treatment for an active AIDS-defining opportunistic infection within 90 days prior to screening.
10. Any history of cardiac rhythm disturbance requiring medical or surgical therapy.
11. Any history of acute or chronic pancreatitis.
12. Use of the following medications that carry risk of torsades de pointes: amiodarone, arsenic trioxide, astemizole, bepridil, chloroquine, chlorpromazine, cisapride, clarithromycin, disopyramide, dofetilide, domperidone, droperidol, erythromycin, halofantrine, haloperidol, ibutilide, levomethadyl, mesoridazine, methadone, pentamidine, pimozide, probucol, procainamide, quinidine, sotalol, sparfloxacin, terfenadine, thioridazine.
13. Receipt of compounds with HDAC inhibitor-like activity, such as valproic acid within the last 30 days. Potential participants may enroll after a 30-day washout period.
14. Known hypersensitivity to the components of VOR or its analogs.
15. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
16. Pregnancy or breast feeding, or expecting to father children within the projected duration of the study.
17. Inability to communicate effectively with study personnel.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-02; Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Margolis, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Archin NM, Liberty AL, Kashuba AD, Choudhary SK, Kuruc JD, Crooks AM, Parker DC, Anderson EM, Kearney MF, Strain MC, Richman DD, Hudgens MG, Bosch RJ, Coffin JM, Eron JJ, Hazuda DJ, Margolis DM. Administration of vorinostat disrupts HIV-1 latency in patients on antiretroviral therapy. Nature. 2012 Jul 25;487(7408):482-5. doi: 10.1038/nature11286. PMID 22837004
- [Result] Archin NM, Bateson R, Tripathy MK, Crooks AM, Yang KH, Dahl NP, Kearney MF, Anderson EM, Coffin JM, Strain MC, Richman DD, Robertson KR, Kashuba AD, Bosch RJ, Hazuda DJ, Kuruc JD, Eron JJ, Margolis DM. HIV-1 expression within resting CD4+ T cells after multiple doses of vorinostat. J Infect Dis. 2014 Sep 1;210(5):728-35. doi: 10.1093/infdis/jiu155. Epub 2014 Mar 11. PMID 24620025
- [Derived] Garrido C, Tolstrup M, Sogaard OS, Rasmussen TA, Allard B, Soriano-Sarabia N, Archin NM, Margolis DM. In-vivo administration of histone deacetylase inhibitors does not impair natural killer cell function in HIV+ individuals. AIDS. 2019 Mar 15;33(4):605-613. doi: 10.1097/QAD.0000000000002112. PMID 30830886
- [Derived] Archin NM, Kirchherr JL, Sung JA, Clutton G, Sholtis K, Xu Y, Allard B, Stuelke E, Kashuba AD, Kuruc JD, Eron J, Gay CL, Goonetilleke N, Margolis DM. Interval dosing with the HDAC inhibitor vorinostat effectively reverses HIV latency. J Clin Invest. 2017 Aug 1;127(8):3126-3135. doi: 10.1172/JCI92684. Epub 2017 Jul 17. PMID 28714868

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential HIV infected participants who were durably suppressed (<50 copies/mL) on stable ART with a CD4 count >300/μL were recruited from the UNC ID clinic and UNC AIDS Clinical Trials Unit. Twenty seven (27) participants were screened for both study periods, 25 unique individuals enrolled between February 2011 and March 31, 2016.
Pre-assignment Details: Participants were recruited into the single and multiple dose Vorinostat (VOR) Arm alone, the VOR Interval Dosing Arm alone, or both = 25. Each Arm had multiple steps. Participants without a significant in vitro or in vivo response to VOR did not advance in either Arm; 3 Arm 1 and 13 new participants, enrolled Arm 2.
Groups:
- Single and Multiple Dose: There are 3 Steps in this Arm: Step 1 a Baseline leukapheresis was completed to obtain resting CD4+ T cells for quantitation of resting CD4+ T cell infection (RCI) and resting CD4+ T cell- associated HIV RNA (RCVL); ex-vivo exposure. Step 2 measured the in-vivo response to single dose of VOR; Step 3 measured the in vivo response after each of 2 series of exposure to multiple doses of VOR 400 mg PO. In each series, 11 doses of VOR were administered for 3 days (M-T-W) and no doses for the remaining 4 days. A leukapheresis was completed 4 hours after the 11th dose to measure in vivo response.
- Interval Dosing: There are 4 steps in this Arm. Step 1 Baseline leukapheresis (Visit 2) to obtain resting CD4+ T cells for quantitation of resting CD4+ T cell infection (RCI) and resting CD4+ T cell- associated HIV RNA (RCVL). Ex-vivo exposure to measure RCVL responsiveness to Vorinostat. Step 2 involved measurement of in vivo response to single dose of VOR. Step 3 involved 2 doses separated by 48 or 72 hours. In vivo responsiveness measured for optimal dose interval and step advancement. Step 4 measured significance of response to VOR 400 mg PO taken every 72 hours for 10 doses.
Period: Overall Study
Arm/Group | Single and Multiple Dose | Interval Dosing
Started | 12 | 13
Step 1 (Demonstrating an ex vivo response to VOR, measured in research lab, permitted study advancement) | 8 | 11 (The 2 participants without an ex vivo response were terminated from the study.)
Step 2 (Demonstrated an in vivo response to a single VOR 400 mg PO in Step 2) | 8 (These participants demonstrated an ex vivo response in Step 1) | 4 (The 7 participants without an in vivo response to single dose of VOR 400 mg PO were terminated.)
Step 2 (Did not demonstrate an in vivo response to VOR 400 mg PO) | 4 (The 4 without ex vivo response (Step 1) took a single dose to see if in vivo response would occur) | 0
Step 3 (Demonstrated an in vivo response to multiple doses of VOR 400 mg PO) | 0 (None who qualified for the 2 series of 11 doses of VOR (taken M-T-W & off for 4 days for 4 wks).) | 6 (3 Arm 1 participants enrolled here; 6/7 had in vivo response to 2 VOR doses given 72 hours apart.)
Step 4 (Demonstrated an in vivo response to 10 doses taken a designated intervals) | 0 (Arm 1 did not have a Step 4) | 3 (Only 3/6 completed the study.)
Completed | 0 | 3
Not Completed | 12 | 10
Not completed — No ex vivo or in vivo response | 4 | 0
Not completed — Physician Decision | 3 | 0
Not completed — Lack of Efficacy | 5 | 9
Not completed — No in vivo response to interval doses | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Single, Multiple and Interval Dosing Of Vorinostat 400 mg PO: The study was separated into Arms for reporting purposes required in this report. The data representing the eligibility and baseline measures were the same throughout the study and are therefore reported as a composite of the entire study. Vorinostat 400 mg PO was administered in single and multiple doses in both Arm 1 and 2. The entire cohort is described below and representative of all who were enrolled in the study over the 5 year period.
Arm/Group | Single, Multiple and Interval Dosing Of Vorinostat 400 mg PO
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 49 [23 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 1
  Black or African American | 4
  Caucasian or White | 20
Region of Enrollment [Number; unit: participants]
  United States | 25
HIV-1 RNA Categories [Count of Participants; unit: Participants]
  < 50 copies/mL | 25
  >= 50 copies/mL | 0
CD4 Nadir [Median (Full Range); unit: cells/µL] | 403 [49 to 879]
CD4 Cell Count [Median (Full Range); unit: cells/µL] | 718 [402 to 1302]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Exhibiting an in Vivo Resting CD4+ T Cell- Associated HIV RNA (RCVL) Increase After Receiving a Single Dose of VOR 400 mg PO
Description: Participants in Arm 1 and 2 were analyzed in Step 2 for an in vivo increase in resting CD4+ T cell- associated HIV RNA (RCVL) after administration of a single dose of VOR 400 mg PO
Time Frame: Arm1: Baseline, Visit 5 and Arm 2: Baseline and Visit 3
Measure: Count of Participants; unit: Participants
Groups:
- 1/Single & Multiple Dose, Step 2, Visit 5: Participants enrolled in Arm 1 were given one dose of VOR 200 mg by mouth (PO), symptoms were assessed over 12 hours and pharmacokinetic samples obtained. Leukapheresis procedure was performed 4 hours after the dose to measure RCVL in-vivo response.
- 2/Interval Dosing, Visit 3: Participants enrolled in Arm 2 receiving a single dose of VOR 400 mg PO after demonstrating an ex vivo response at baseline. Symptoms were assessed over 12 hours and pharmacokinetic samples obtained. Leukapheresis procedure was performed 4 hours after the dose to measure RCVL in-vivo response.
Arm/Group | 1/Single & Multiple Dose, Step 2, Visit 5 | 2/Interval Dosing, Visit 3
Number analyzed (Participants) | 12 | 11
Participants | 8 | 4

2. Primary Outcome: Number of Participants Exhibiting an in Vivo Resting CD4+ T-cell-associated HIV RNA (Rc-RNA) Increase Following Each of Two Multiple Dose Cycles (11 Doses/Cycle)
Description: Participants in Arm 1, Step 3 were analyzed for an in vivo increase in the resting CD4+ T cell- associated HIV RNA (RCVL) after 11 doses of VOR 400 mg PO. This cycle was repeated after a 5 - 8 week rest period for a 2nd series and measurement.
Time Frame: Baseline, Visit 18, Visit 29
Population: Participants with resting CD4+ T-cell-associated HIV RNA (rc-RNA) increases after receiving daily VOR Monday through Wednesday for 8 weekly cycles were enrolled.
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1 - Single and Multiple Dose, Step 3: Participants without dose-limiting symptoms and exhibiting an in vivo response to single VOR doses were eligible to receive multiple doses of VOR 400 mg. The first dose was administered in clinic with observation for symptoms for 1 hour post dose. Symptoms were assessed daily and on the third day 4 hours after the dose. These participants took VOR 400 mg (PO) in the AM for 3 days each week (dose every M-T-W) for 3 weeks. On the 4th week, the participant took 2 doses of VOR 400 mg (M-T) in the AM. A leukapheresis was completed 4 hours after the 2nd dose of VOR to measure RCVL in-vivo response. After a 4 - 8 week rest period, participants without dose-limiting symptoms repeated the 4 week cycle.
Arm/Group | Arm 1 - Single and Multiple Dose, Step 3
Number analyzed (Participants) | 5
Participants | 0

3. Primary Outcome: Number of Participants With a Significant in Vivo Response in Resting Cell Infection (RCI) and HIV RNA After Paired Doses
Description: Induction of significant in vivo RCI and RCLV response after 2 doses of VOR 400 mg PO administered 48 hours apart or 72 hours apart
Time Frame: Baseline, Visit 6
Population: Participants showing an in vivo response in resting CD4+ T cell- associated HIV RNA (RCVL) after a single dose of VOR were administered 2 doses of VOR 400 mg separated by either 48 or 72 hours to determine the optimal interval/spacing to observe a significant in vivo response in the RCVL after the paired doses.
Measure: Count of Participants; unit: Participants
Groups:
- Interval Dosing , Step 3 (48 hr Interval): Participants without dose-limiting symptoms and exhibiting an in vivo response to single VOR dose were eligible to receive 2 doses of VOR 400 mg PO, given at the pre-determined interval of 48 hours. Participant took the PO doses at home per schedule with daily telephone assessment of symptoms. Leukapheresis procedure performed 4 hours after the 2nd dose to measure RCVL in-vivo response.
- Interval Dosing, Step 3 (72 Hour Interval): Participants without dose-limiting symptoms and exhibiting an in vivo response to single VOR dose were eligible to receive 2 doses of VOR 400 mg PO, given at the pre-determined interval of 72 hours. Participant took the PO doses at home per schedule with daily telephone assessment of symptoms. Leukapheresis procedure performed 4 hours after the 2nd dose to measure RCVL in-vivo response.
Arm/Group | Interval Dosing , Step 3 (48 hr Interval) | Interval Dosing, Step 3 (72 Hour Interval)
Number analyzed (Participants) | 1 | 7
Participants | 0 | 6

4. Primary Outcome: Number of Participants Exhibiting an in Vivo Resting CD4+ T-cell-associated HIV RNA (Rc-RNA) Increase Following Multiple (n = 10) Interval Doses
Description: Participants in Arm 2, Step 4 were analyzed for an in vivo increase in the resting CD4+ T cell- associated HIV RNA (RCVL) after administration of 10 doses of VOR 400 mg PO, given 72 hours apart.
Time Frame: Baseline, Visit 9
Population: Participants who demonstrated a significant in vivo response after taking 2 doses of VOR 400 mg PO, each dose taken 72 hours apart were administered 10 doses of VOR based on the optimal dosing of 72 hours.
Measure: Count of Participants; unit: Participants
Groups:
- Interval Doses (Multiple) Step 4: Participants without dose-limiting symptoms and exhibiting an in vivo response to the paired doses of VOR 400 mg PO were eligible to receive 10 doses of VOR, given at the pre-determined interval. Participant took the PO doses at home per schedule with daily telephone assessment of symptoms and clinical assessments at after the 3rd, 5th, 8th and 10th doses. Participant were only given the required doses for administration between visits.
  Leukapheresis procedure performed 4 hours after the 10th dose to measure RCVL in-vivo response.
Arm/Group | Interval Doses (Multiple) Step 4
Number analyzed (Participants) | 3
Participants | 3

5. Secondary Outcome: Number of Participants With Measurable Changes in Plasma HIV-1 RNA
Description: Assess for detectible HIV-1 RNA > 150 copies/mL, confirmed by repeat evaluation, following VOR dose. By standard assay and single copy assay. Pre specified to combine all participants into one arm.
Time Frame: 1 week after last VOR dose
Population: All participants receiving one or more doses of VOR in any and all Arms of the study.
Measure: Count of Participants; unit: Participants
Groups:
- 1/Single & Multiple Dose, Steps 2 and 3: All eligible participants in the Single and Multiple Group Arm who received at least one dose of VOR 400 mg PO
- 2/Interval Dosing, Steps 2, 3 and 4: All eligible participants in the Interval Dosing Arm who received at least one dose of VOR 400 mg PO
Arm/Group | 1/Single & Multiple Dose, Steps 2 and 3 | 2/Interval Dosing, Steps 2, 3 and 4
Number analyzed (Participants) | 12 | 13
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With Confirmed Non-hematologic Toxicity >/= Grade 3 and Related to VOR Per Division of AIDS (DAIDS) Grading Table
Description: DAIDS Grading Table- Grade 1- mild, Grade 2- moderate; Grade 3- severe Grade 4- potentially life-threatening. Pre specified to combine all participants into one arm.
Time Frame: 24 hrs following single dose and 1 week after last of multiple dose sequence
Population: All participants receiving one or more doses of VOR 400 mg PO in any and all Arms of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Single & Multiple Dose, Steps 2 and 3 | 2/Interval Dosing, Steps 2, 3 and 4
Number analyzed (Participants) | 12 | 13
Participants | 0 | 0

7. Secondary Outcome: Number of Participants With Confirmed Hematologic Toxicity >/= Grade 2 and Related to VOR Per Division of AIDS (DAIDS) Grading Table
Description: as for outcome 6
Time Frame: 24 hrs following single dose and 1 week after last of multiple dose sequence
Population: All participants receiving one or more doses of VOR 400 mg PO in any and all Arms of the study.
Measure: Count of Participants; unit: Participants
Groups:
- 1/Single & Multiple Dose, Steps 2 and 3: All eligible participants in the Single and Multiple Arm who received at least one dose of VOR 400 mg PO.
Arm/Group | 1/Single & Multiple Dose, Steps 2 and 3 | 2/Interval Dosing, Steps 2, 3 and 4
Number analyzed (Participants) | 12 | 13
Participants | 0 | 0

8. Other Pre Specified Outcome: Number of Participants Developing Cancer Within 5 Years Following >/= 8 Vorinostat Dose Exposures
Description: Development of a new cancer within the 5 years of taking their last dose of VOR 400 mg PO.All participants receiving one or more doses of VOR 400 mg PO in any and all Arms of the study. Pre-specified to be reported as one group.
Time Frame: From last dose Vorinostat to 5 years afterwards
Population: At end of study, participants receiving >/= 8 doses of Vorinostat are enrolled in a 5-year cancer incidence database to be monitored for the occurrence of cancer.
Measure: Count of Participants; unit: Participants
Groups:
- 1/Single and Multiple Dose, Step 3: Participants without dose-limiting symptoms and exhibiting an in vivo response to single VOR doses were eligible to receive multiple doses of VOR 400 mg. The first dose was administered in clinic with observation for symptoms for 1 hour post dose. Symptoms were assessed daily and on the third day 4 hours after the dose. These participants took VOR 400 mg (PO) in the AM for 3 days each week (dose every M-T-W) for 3 weeks. On the 4th week, the participant took 2 doses of VOR 400 mg (M-T) in the AM. A leukapheresis was completed 4 hours after the 2nd dose of VOR to measure RCVL in-vivo response. After a 4 - 8 week rest period, participants without dose-limiting symptoms repeated the 4 week cycle.
- 2/Interval Doses (Multiple) Step 4: Participants without dose-limiting symptoms and exhibiting an in vivo response to the paired dose of VOR dose were eligible to receive 10 doses of VOR 400 mg PO, given at the pre-determined interval. Participant took the PO doses at home per schedule with daily telephone assessment of symptoms and clinical assessments at after the 3rd, 5th, 8th and 10th doses. Participant were only given the required doses for administration between visits.
  Leukapheresis procedure performed 4 hours after the 10th dose to measure RCVL in-vivo response.
Arm/Group | 1/Single and Multiple Dose, Step 3 | 2/Interval Doses (Multiple) Step 4
Number analyzed (Participants) | 5 | 3
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Period One: February 1, 2011 through December 31, 2013. Period Two: January 1, 2014 through March 31, 2016.
Description: Data were analyzed for all participants in one arm.
Groups:
- Open Label - Translational Research Study: Period One: Step 1 (ex-vivo), Step 2 (single dose) and Step 3 (multiple dose). Advancement to each step required demonstration of significant HIV-1 RNA expression per 1 million RCVL response to VOR. Step 1: All participants had an ex-vivo exposure to VOR. Step 2: Participants with and without an ex-vivo response received 1 single dose VOR. Step 3: Participants demonstrating an in vivo response received multiple doses consisting of 2 series of 11 VOR doses each; with in vivo response measured after each series. Period One was stopped due to lack of significant in-vivo response to the multiple doses.
  Period Two: Step 1, Step 2 and advancement criteria are the same as above. Step 3 (interval paired dose) and Step 4 (multiple interval doses). Participants without an ex-vivo response did not progress past Step 1. Step 3: Responders received 2 doses separated by 48 or 72 hours. Step 4: Responders then received 10 doses of VOR at pre-determined interval.
Arm/Group | Open Label - Translational Research Study
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 21/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label - Translational Research Study (N=25)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (2)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Blood Albumin Decreased (Investigations) | 2 (2)
Blood Calcium Decreased (Investigations) | 1 (1)
Blood Calcium Increased (Investigations) | 1 (1)
Blood Creatinine Increased (Investigations) | 2 (3)
Blood Glucose Increased (Investigations) | 9 (16)
Blood Potassium Decreased (Investigations) | 3 (3)
Blood Sodium Increased (Investigations) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (3)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Dizziness (Nervous system disorders) | 6 (8)
Dizziness Postural (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Euphoric Mood (Psychiatric disorders) | 1 (1)
Fatigue (General disorders) | 7 (9)
Haemoglobin Decreased (Investigations) | 1 (2)
Headache (Nervous system disorders) | 5 (10)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1)
Memory Impairment (Nervous system disorders) | 1 (1)
Mental Impairment (Nervous system disorders) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (13)
Neutrophil Count Decreased (Investigations) | 2 (4)
Night Sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Pallor (Vascular disorders) | 1 (1)
Platelet Count Decreased (Investigations) | 3 (5)
Post Procedural Hematoma (Injury, poisoning and procedural complications) | 2 (2)
Post Procedural Oedema (Injury, poisoning and procedural complications) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Procedural Anxiety (Injury, poisoning and procedural complications) | 1 (1)
Procedural Complication (Injury, poisoning and procedural complications) | 1 (1)
Procedural Dizziness (Injury, poisoning and procedural complications) | 1 (1)
Procedural Headache (Injury, poisoning and procedural complications) | 2 (2)
Procedural Hypertension (Injury, poisoning and procedural complications) | 17 (44)
Procedural Nausea (Injury, poisoning and procedural complications) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 2 (2)
Procedural Site Reaction (Injury, poisoning and procedural complications) | 9 (15)
Thirst (General disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Vascular Access Site Haematoma (Injury, poisoning and procedural complications) | 4 (4)
Vascular Access Site Haemorrhage (Injury, poisoning and procedural complications) | 6 (7)
Vascular Access Site Pain (Injury, poisoning and procedural complications) | 8 (8)
Vascular Access Site Rupture (Injury, poisoning and procedural complications) | 4 (5)
Vascular Access Site Swelling (Injury, poisoning and procedural complications) | 4 (4)
Vessel Puncture Site Erythema (General disorders) | 1 (1)
Vessel Puncture Site Haematoma (General disorders) | 1 (1)
Visual Impairment (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No